CLINICAL TRIAL: NCT06517888
Title: A Phase 1/2 Trial of AAVAnc80-antiVEGF Gene Therapy in Individuals With Unilateral Vestibular Schwannoma
Brief Title: Anti-VEGF Gene Therapy Trial for Vestibular Schwannoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akouos, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK-antiVEGF-101
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular schwannoma; Hearing loss; Acoustic neuroma; anti-VEGF
MeSH Terms: conditions — Neuroma, Acoustic; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Adult participants to receive a single unilateral intracochlear administration of AAVAnc80-antiVEGF (dose level 1) in the study ear using a sterile, one-time use investigational medical device.
  Interventions: Combination Product: AAVAnc80-antiVEGF via Akouos Delivery Device
- Cohort 2 (Experimental): Adult participants to receive a single unilateral intracochlear administration of AAVAnc80-antiVEGF (dose level 2) in the study ear using a sterile, one-time use investigational medical device.
  Interventions: Combination Product: AAVAnc80-antiVEGF via Akouos Delivery Device
- Cohort 3 (Experimental): Adult participants to receive a single unilateral intracochlear administration of AAVAnc80-antiVEGF (dose level 3) in the study ear using a sterile, one-time use investigational medical device
  Interventions: Combination Product: AAVAnc80-antiVEGF via Akouos Delivery Device

INTERVENTIONS:
Combination Product: AAVAnc80-antiVEGF via Akouos Delivery Device — AAVAnc80-antiVEGF is a sterile suspension intended to be administered via intracochlear administration as a single dose using the Akouos Delivery Device

SUMMARY:
This trial will evaluate the safety and tolerability of a single unilateral administration of one of three dose levels of AAVAnc80-antiVEGF and will evaluate the Akouos delivery device to safely achieve the intended product performance.

ELIGIBILITY:
Criteria for Inclusion:

1. Presence of unilateral, progressive vestibular schwannoma.
2. Vestibular schwannoma larger than 2 mm.
3. Profound hearing loss, defined by pure-tone audiometry thresholds or word recognition score, in the affected ear.
4. Able and willing to comply with all trial requirements, including willingness to participate in a separate long term follow-up study after completion of this trial.

Criteria for Exclusion:

1. Prior diagnosis of NF2 and/or bilateral vestibular schwannoma.
2. Prior surgery or radiation therapy for vestibular schwannoma.
3. Clinical history consistent with endolymphatic hydrops (documented fluctuating sensorineural hearing loss and/or episodic vertigo) in the affected ear.
4. Profound hearing loss, defined by pure-tone audiometry thresholds or word recognition score, in the unaffected ear.
5. Prior participation in a clinical trial with an investigational drug within six months prior to administration (Day 0), or any prior participation in a gene therapy clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | through trial completion, approximately one year
  AEs with relationship to the investigational medicinal product and/or to the administration procedure (including the delivery device)

SECONDARY OUTCOMES:
Tumor Volume | through trial completion, approximately one year
  Change from baseline in tumor size via MRI (volumetric analysis)
Performance of Akouos Delivery Device | through trial completion, approximately one year
  Performance based on the frequency of device deficiencies observed during delivery of AAVAnc80-antiVEGF to the intracochlear space

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Reape, MD, Study Director — Akouos, Inc.
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt Bill Wilkerson Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No